CLINICAL TRIAL: NCT04875572
Title: Association of Analgesia Nociceptive Index With Preoperative Anxiety: A Prospective Observational Study
Brief Title: Associations Between Analgesia Nociception Index and Preoperative Anxiety
Acronym: PANIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Anthony Chau, Principle Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H19-03148
Record Dates: First submitted 2021-02-23; First posted 2021-05-06 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Anxiety; Opioid Consumption; Cesarean Section
Keywords: Analgesia Nociception Index; Prospective Observational Study
MeSH Terms: conditions — Anxiety Disorders | interventions — Monitoring, Physiologic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Since this is a single group study, all patients enrolled will receive the same care, as described in the study description above.
  Interventions: Device: Analgesia Nociception Index (ANI) Monitor

INTERVENTIONS:
Device: Analgesia Nociception Index (ANI) Monitor — The ANI monitor produces an objective measure of parasympathetic tone through non-invasive electrodes placed on the patient's chest. The patient's standard of care is not affected, and the anesthetist is blinded to the monitor, so as not to affect their anesthetic practice.

SUMMARY:
The management and prediction of pain is one of the most crucial jobs for anesthetists. It has been shown that a patient's ability to remain calm during stressful situations is related to their post-surgical pain scores. The MetroDoloris Analgesia Nociception Index (ANI) monitor is a heart-rate monitor that provides us with a number which reflects a patient's state of relaxation (or parasympathetic tone). For this reason, the investigators are testing whether ANI can be used as a metric for perioperative anxiety, and a predictive tool for pain after c-sections.

DETAILED DESCRIPTION:
Purpose: The purpose of the study is to evaluate the MDoloris ANI monitor as an effective tool for objectively measuring perioperative stress, and as a prediction of post-operative pain.

Hypothesis: High perioperative anxiety scores, high post-operative pain scores, high post-operative anesthetic dosing, and high incidence of provider intervention will be positively correlated with frequency and magnitude of changes in the ANI score.

Justification: Anesthetists are constantly monitoring a patient's heart rate during caesarean sections. This is standard care, and this monitoring provides useful information about a patient's level of sedation, analgesia, and comfort. The ANI monitor takes more heart rate information through two electrodes placed on a patient's chest, and non-invasively provides more information by which anesthetists can improve the patient's standard of care.

Primary Objective: To determine whether the ANI monitor is a viable means of measuring perioperative anxiety during C-sections.

Secondary Objectives:

To determine if the ANI monitor is capable of providing anesthetists with an objective prediction variable for post-operative pain.

Research Methods and Design: Once eligibility is determined , the patient will be approached in the pre-operative waiting area at a time determined by the charge nurse. If they consent to the study, they will be given an validated questionnaire which assesses the patient's level of operative stress. After the survey, they will have the ANI electrodes placed on their chest by a member of the study team. The collection of this pre-surgical data provides the research team with a baseline to which they will compare the operative and post-operative results. Five to ten minutes prior to their surgery, the electrodes will be removed, and the monitor will be brought to the OR. The monitor will be plugged in to an electrical socket far away from areas of high traffic, and will not disturb the flow of OR staff.

During the operation, a member of the study team will constantly watch the ANI monitor to check for optimal connectivity, and will record the events of surgery. A record of the events is critical to interpreting the meaning of the ANI score, as it allows the team to match distinct stimuli with the number produced by the monitor.

The spinal block typically wears off after 24 hours, so at 24- and 48 hours following the c-section, a study team member will approach the patient on the wards, and ask for their resting, and evoked pain scores on a VAS 0-100 mm scale. Evoked pain is pain caused by movement. The investigators have chosen the previously used metric of a change in position: from lying to sitting. If the patient has received drugs for pain already, the investigator will ask them to score the pain they experienced before receiving medication. The study investigator will finally record the provider-administered dose of pain medication from the patient's chart.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older.
* Patient receiving an uncomplicated, scheduled caesarean section
* Patient with a normal sinus rhythm

Exclusion Criteria:

* Presentation with cardiac arrhythmia
* Contraindications to neuraxial analgesia (ex. patient refusal, infection at the site of injection, uncorrected hypovolemia, allergy, increased intracranial pressure, coagulopathy, sepsis, fixed cardiac output states, or indeterminate neurological status), or risk factors likely to affect placement or function of the spinal needle (ex. previous back surgery, significant uncorrected scoliosis, or morbid obesity (BMI >40))
* History of hypersensitivity or idiosyncratic reaction to local anesthetics or opioids
* Current or historical evidence of any significant medical conditions, including diseases of pregnancy
* Clinical settings in which general anesthesia may be preferable (ex. patient with failed regional anesthetic, patient with history of bleeding, fetal shoulder dystocia etc.)
* Anticipated fetal abnormalities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Validation of Analgesia Nociception Index (ANI) score for objective measurement of anxiety | 25 minutes perioperatively
  Association between frequency and magnitude of changes in ANI during the perioperative time period with patient's reported perioperative anxiety scores
Validation of ANI score for prediction of post-operative pain 24 hours | Pain scores at 24 hours
  Association between frequency and magnitude of changes in the ANI with patient's reported VAS evoked and resting pain scores at 24h and 48h. Evoked pain is defined as pain experienced from moving from a supine position (where resting pain VAS is measured) to seated position.
Validation of ANI score for prediction of post-operative pain 48 hours | Pain scores at 48 hours
  Association between frequency and magnitude of changes in the ANI with patient's reported VAS evoked and resting pain scores at 24h and 48h. Evoked pain is defined as pain experienced from moving from a supine position (where resting pain VAS is measured) to seated position.

SECONDARY OUTCOMES:
Validation of ANI score for prediction of post-operative opioid requirements at 24 hours | Opioid use collected during followup at 24 hours
  Association between frequency and magnitude of changes in the ANI with patient's total opioid consumption in oral morphine equivalents at 24h and 48h
Validation of ANI score for prediction of post-operative opioid requirements at 48 hours | Opioid use collected during followup at 48 hours
  Association between frequency and magnitude of changes in the ANI with patient's total opioid consumption in oral morphine equivalents at 24h and 48h
Absolute ANI score validation at 24 hours | Pain score recorded 24 hours post partum
  Determining whether post-partum pain, and operative anxiety are correlated with frequency of absolute ANI score less than 50
Absolute ANI score validation at 48 hours | Pain score recorded at 48 hours post partum
  Determining whether post-partum pain, and operative anxiety are correlated with frequency of absolute ANI score less than 50
Percent variability in ANI | ANI score recorded for 25 minutes perioperatively
  Use of Percent Variability (PV) statistic as a measure of top-down regulation of parasympathetic tone

CONTACTS AND LOCATIONS:
Overall Officials: Anton Chau, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada

DOCUMENTS (2):
  • Study Protocol (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT04875572/Prot_000.pdf
  • Informed Consent Form (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT04875572/ICF_001.pdf